CLINICAL TRIAL: NCT01046214
Title: A Multiple-Dose, Double Blind, Double Dummy, Comparative Bioavailability Study of Two Formulations of Bupropion Hydrochloride 300 mg Extended Release Tablets Under Fasting Conditions
Brief Title: Bupropion Hydrochloride 300 mg Extended Release Tablets Under Fasting Conditions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2008-1668
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budeprion XL™ (Experimental): Budeprion XL™ 300 mg Extended Release Tablet dosed once daily for 8 days, in the morning, after an overnight fast of at least 10 hours, with the reference-placebo tablet
  Interventions: Drug: Bupropion HCl
- Wellbutrin XL® (Active Comparator): Wellbutrin XL® 300 mg Extended Release Tablet dosed once daily for 8 days, in the morning, after an overnight fast of at least 10 hours, with the test-placebo tablet
  Interventions: Drug: Bupropion HCl

INTERVENTIONS:
Drug: Bupropion HCl — Budeprion XL™ 300 mg Extended Release Tablet dosed once daily for 8 days, in the morning, after an overnight fast of at least 10 hours, with the reference-placebo tablet
  Other Names: Budeprion XL™
  Arms: Budeprion XL™
Drug: Bupropion HCl — Wellbutrin XL® 300 mg Extended Release Tablet dosed once daily for 8 days, in the morning, after an overnight fast of at least 10 hours, with the test-placebo tablet
  Other Names: Wellbutrin XL®
  Arms: Wellbutrin XL®

SUMMARY:
The objective of this study is to evaluate the comparative bioavailability between bupropion hydrochloride 300 mg extended release tablets (Teva Pharmaceuticals USA) and Wellbutrin XL® 300 mg extended release tablets (Biovail Pharmaceuticals, Inc.) at steady-state in patients under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 25 years of age or older
* Diagnosis of any depressive disorder as per DSM IV criteria (except bipolar depression and major depressive disorder with psychotic features). Note: Both patients who are or are not being treated with bupropion or other antidepressants are permitted into the study.
* Patients must have complained of suffering from adverse events and/or lack of effect when switched from Wellbutrin XL® 300 mg to Budeprion XL™ 300 mg.
* BMI (kg/m2) Greater than or equal to 19 and less than or equal to 34.
* No clinically significant abnormal laboratory values
* No clinically significant findings in a 12-lead electrocardiogram (ECG)
* No clinically significant findings in vital signs measurements.
* Be informed of the nature of the study and give written consent prior to receiving any study procedure.

Exclusion Criteria

* Carcinoma within the last 5 years. Note: Patients with basal or squamous cell carcinoma may be permitted into the study on a case by case basis.
* A history of epilepsy or risk for seizures.
* A previous or current diagnosis of bipolar depression.
* A current diagnosis of major depressive episode with psychotic features. Note: Subjects with previous diagnosis of major depressive episode with psychotic features may be included at the investigator's discretion.
* A previous or current diagnosis of an eating disorder (e.g. bulimia, anorexia nervosa).
* A lifetime history of schizophrenia or schizo-affective disorder.
* Significant disease(s) or clinically significant finding(s) in a physical examination determined by an investigator to pose a health concern to the patient while on study.
* Presence of clinically significant gastrointestinal disease and/or surgery (e.g. gastric bypass surgery) or history of malabsorption within the last year.
* Known history or presence of an allergic sensitivity to bupropion and/or any other drug substances with similar activity.
* Expected changes in use of permitted concomitant medication that will be continued throughout the study.
* Undergoing abrupt discontinuation of sedatives (including benzodiazepines).
* Use of monoamine oxidase inhibitors (MAOI) within 2 weeks prior to study admission.
* Taking medications that interact with CYP2B6 within 30 days prior to Day 1 dosing.
* Taking levodopa, amantadine, drugs that lower seizure threshold (e.g. theophylline, systemic steroids, antipsychotics), and/or on nicotine replacement therapy.
* History of alcohol or drug-dependence by DSM IV criteria within 6 months prior to study admission.
* Positive test results for:

  * HIV
  * Hepatitis B surface antigen or Hepatitis C antibody
  * Urine drugs of abuse (i.e. marijuana, amphetamines, barbiturates, cocaine, opiates, methadone, and phencyclidine) Note: any positive test result(s) for benzodiazepine(s) must be assessed by the investigator to determine whether the patient should be excluded from this study.
  * Serum hCG consistent with pregnancy (females only).
* On a special diet within 30 days prior to study admission (e.g. liquid, protein, raw food diet).
* Difficulty fasting or consuming standard meals.
* Participated in another clinical trial or received an investigational product within 45 days prior to Day 1 drug administration.
* Donation or loss of whole blood:

  * Less than or equal to 499 mL within 30 days prior to dosing
  * Greater than or equal to 500 mL within 56 days prior to dosing Note: blood taken for routine medical evaluations totaling less than 50 mL will be permitted.
* Females who have discontinued the use of:

  * implanted, intrauterine, or injected hormonal contraceptives within 6 months prior to Day 1 drug administration, OR
  * oral, intravaginal, or patch hormonal contraceptives within 1 month prior to Day 1 drug administration
* Females who started taking:

  * implanted or intrauterine hormonal contraceptives less than 6 months prior to Day 1 drug administration, OR
  * oral, intravaginal, patch, or injected hormonal contraceptives less than 3 months prior to Day 1 drug administration.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Have had a newly applied tattoo or body piercing within 30 days prior to study admission.
* Does not tolerate venipuncture.
* Unable or unwilling to provide informed consent.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01

PRIMARY OUTCOMES:
Comparative bioavailability | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lev Gertsik, MD, Principal Investigator — California Clinical Trials
Locations (2):
- United States (2):
  - California Clinical Trials, Culver City, California
  - California Clinical Trials, Glendale, California